CLINICAL TRIAL: NCT06157593
Title: Neurally Adjusted Ventilatory Assist for Weaning From Invasive Mechanical Ventilation in Critically Ill Children: A Randomised Control Trial
Brief Title: Neurally Adjusted Ventilatory Assist for Weaning From Invasive Mechanical Ventilation in Critically Ill Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chulalongkorn University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 24112566
Record Dates: First submitted 2023-11-24; First posted 2023-12-06 (Actual); Last update posted 2023-12-06 (Actual); Status verified 2023-11

CONDITIONS: Mechanical Ventilator Weaning; Critically Ill; Mechanical Ventilation; Neurally Adjusted Ventilatory Assist
MeSH Terms: conditions — Critical Illness

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- NAVA (Experimental)
  Interventions: Procedure: NAVA
- SIMV (No Intervention)

INTERVENTIONS:
Procedure: NAVA — weaning from mechanical ventilator using neurally adjusted ventilatory assist
  Arms: NAVA

SUMMARY:
The goal of this clinical trial is to compare weaning from mechanical ventilation in critically ill children. The main questions it aims to answer are:

* Will weaning with neurally adjusted ventilatory assist (NAVA) mode ventilation result in shorter ventilator day than synchronised intermittent mandatory ventilation (SIMV) mode?
* Will weaning with NAVA mode ventilation result in shorter paediatric intensive care unit (PICU) length of stay than SIMV mode? Participants will be randomised to NAVA or SIMV group for weaning from mechanical ventilation, then PICU outcomes from both groups will be collected, analysed and compared.

ELIGIBILITY:
Inclusion Criteria:

* all critically ill children admitted to PICU

Exclusion Criteria:

* failure to obtain informed consent

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-02 (Estimated); Primary Completion 2025-02 (Estimated); Study Completion 2025-07 (Estimated)

PRIMARY OUTCOMES:
ventilator day | immediately after extubation
  number of days patients receive mechanical ventilation
PICU length of stay | immediately after PICU discharge
  number of days patients remain in PICU

SECONDARY OUTCOMES:
asynchrony index | 20-minute period randomly captured from the day of extubation
  asynchronous breaths divided by total breaths in 20 minutes

CONTACTS AND LOCATIONS:
Locations (1):
- Chulalongkorn University, Bangkok, Thailand

IPD SHARING:
Plan to Share IPD: No